CLINICAL TRIAL: NCT02194868
Title: Role and Interactions Between Immunoregulatory T Lymphocytes Subtypes After Allogeneic Haematopoietic Stem Cell Transplantation (HSCT): Identification of New Partners Implicated on the Development of GVT (Graft Versus Tumor) and Anti-infectious Responses Without GVHD (Graft Versus Host Disease)
Brief Title: Immunoregulatory T Lymphocytes Subtypes and Haematopoietic Stem Cell Transplantation (HSCT)
Acronym: REG-Allo
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI 12036
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation for Hematological Malignancies
Keywords: Allogeneic hematopoietic stem cell transplantation,; Immunoregulatory T lymphocytes,; acute graft versus host disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, hematopoietic stem cell of bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- donors of hematopoietic stem: Adult and minor donors of hematopoietic stem
- patients requiring allogeneic hema: Adult and minor patients (recipients) requiring allogeneic hema
  Interventions: Biological: Recipients

INTERVENTIONS:
Biological: Recipients — 1. Adult recipient:
     * collected 20 ml pre-transplant
     * collected 30 ml for adults on day 20 post-transplant at engraftment for cell phenotype,
     * collected 30 ml on days 30, 60, 90, 180, 360 days post-HSCT for cell phenotyping at all time points, functional INKT at day 60 or 90 depending on the number of cells collected and anti-viral ELISPOT studies on days 180 and 360
  2. Children recipients
     * collected residual blood pre-transplant
     * collected residual blood on day 20 post-transplant at engraftment for cell phenotype,
     * collected residual blood on days 20, 30, 90, 180 and 360 post-HSCT
  Groups: patients requiring allogeneic hema
Biological: Donors — 1. Adult donors :
     * collected 20 ml of blood, (if possible before granulocyte colony-stimulating factor (GCSF) administration)
     * collected 1 ml of the stem cell graft for adult recipient or 2 ml of bone marrow for children recipients These samples will be collected at the same time of those needed for transplant.
  2. Children donors samples
     * collected residual blood
     * 2ml of bone marrow (bottom of tube)

SUMMARY:
The purpose of this study is to confirm that invariant NKT lymphocytes (iNKT) reconstitution in recipient and in the graft content can predict the outcome of human allogeneic HSCT and to set up an algorithm for clinical practice that would allow the prediction of acute GVHD risk according to the quantity and functionality

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) remains the only curative treatment in most haematological malignancies. However, its anti-tumor effect (GVT) is often associated with the development of a graft versus host disease (GVHD) and impaired immune anti-infectious responses. The predictive and protective features of iNKT cells on the development of acute GVHD (aGVHD) are not or poorly known in humans and their mechanisms of action, in particular their potential interactions with the other regulatory effectors and immune actors of the allogeneic response, remain to be explored.

Our project aims, first, to show that the post-transplant reconstitution and/or the content of the graft in some immunoregulatory T lymphocytes can early predict the post-transplant clinical outcome and, second, to explore the underlying immunological mechanisms. For that, we propose to analyse, in homogeneous cohorts of allografted patients and their donors, the levels of iNKT cells and other cell populations implicated in the allogeneic immune response (Tregs, mucosa-associated invariant T (MAIT) cells, delta gammaT and anti-viral specific T cells) and correlate the results to the post-transplant outcome (GVHD, infections, relapse, survival). This study will be performed in a cohort of 80 adult allografted patients in four transplant departments in Paris (hospitals of Necker, Saint Antoine, Saint Louis and La Pitié Salpétrière) and in a cohort of 60 allografted paediatric patients (Robert Debré hospital in Paris). Sequential blood samples of patients will be drawn to monitor the immune reconstitution of the different lymphocyte populations of interest by flow cytometry and perform functional studies on iNKT (ex vivo expansion capacities and cytokine production). These analyses will be also performed in the corresponding donors from blood samples collected before the collection process and from the grafts (obtained by the cell therapy departments of Necker, La Pitié Salpétrière and Saint Louis hospitals). In addition, we plan to analyse the effect of, and the mechanisms by which, human cluster of differentiation 4 (CD4) CD4- and CD4+ iNKT cells might control the allogeneic response in vitro, particularly via their potential interactions with dendritic cells and Tregs. According to the results of the mechanistic studies, we will test the effect of human subtypes of iNKT cells on the GVH/GVL affects in a preclinical humanized mouse model of allogeneic HSCT.

The clinical and biological data will be anonymously entered in the electronic case report by the investigators up to 3 years post transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria for adults:

   * Allogeneic HSCT with peripheral blood stem cell (PBSC) graft
   * Patients transplanted in cytologic Complete Remission (CR)
   * HLA 10/10 on HLA A, B, Cw, DRB1 and DQ molecules, from an intrafamilial or an unrelated donor
   * - Fludarabine-ivBusulfan-ATG based reduced intensity/toxicity conditioning. Iv Busulfan doses between 6.4 mg/kg to 9.6 mg/kg or Fludarabine - TBI ≤ 8 Gy are accepted. ATG should be thymoglobuline at 5 mg/kg
   * Consent form signed by the patient
   * Consent form signed by the donor
   * Affiliated or beneficiary of a health insurance regimen
2. Criteria for pediatric patients:

   * Allogeneic HSCT with bone marrow grafts
   * Myeloablative conditioning (either TBI 12 Gy with Cyclophosphamide or iv Busulfan (12.8 mg/kg) and cyclophosphamide or Fludarabine - TBI > 8 Gy)- HLA 10/10 on HLA A, B, Cw, DRB1 and DQ molecules, from an intrafamilial or an unrelated donor
   * Consent form signed by the parents
   * Consent form signed by the donor or his legal representative if it is minor
   * Beneficiary of a health insurance regimen

Exclusion Criteria:

* History of previous autologous or allogeneic haematopoietic stem cell transplantation
* Disease non in cytologic CR at transplant
* Other type of conditioning than Fludarabine-ivBusulfan-ATG based reduced intensity/toxicity.
* Donor graft with any HLA mismatch including haploidentical and cord blood grafts
* Graft having one or more mismatch with the recipient HLA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The eligible patients will be select by the responsible physicians from clinical teams involved in this study at their BMT staff. These physicians will propose the study to selected patients and provide the informed consent.
  Grafts and blood from donors of patients involved in this study will be provided by the different cell therapy departments related to the clinical groups.
  Peripheral blood from healthy donors will be obtained from volunteer donations to the "Etablissement Français du Sang" (EFS).
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Occurrence of aGVHD | until 3 years post graft
  Patients' clinical files

SECONDARY OUTCOMES:
iNKT and effectors of the immune allogeneic response | until 3 years post graft
  Correlation between iNKT and regulatory effectors of the immune allogeneic response (Assessed by multiparametric flow cytometry of blood sample)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Thérèse Rubio, MD, PhD, Principal Investigator — CHU NANCY; Olivier Hermine, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker, Paris, France